CLINICAL TRIAL: NCT04786938
Title: Effect of Saccaromyces Boulardii CNCM I-745 Supplementation on the Fecal Resistome of Patients Treated Against Helicobacter Pylori Infection
Brief Title: Effect of Probiotics on the Fecal Resistome During Helicobacter Pylori Eradication Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad San Francisco de Quito (Other)
Collaborators: Universidad Tecnológica Equinoccial (Other); Biocodex (Industry)
Responsible Party: Principal Investigator, Paúl Cárdenas, PhD, Professor at the Institute of Microbiology, Universidad San Francisco de Quito
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16943
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Gut Resistome
Keywords: Saccharomyces boulardii; eradication therapy; Helicobacter Pylori [H. Pylori]
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: A total of 72 H. pylori-positive patients were enrolled, and they were randomly assigned to group conventional (A) and group conventional plus S. boulardi (B). Patients in group A received 14-day triple therapy consisting of amoxicillin 1 g three times a day, tinidazole 1 g once a day, and omeprazole 40 mg twice a day. Patients in group B received triple therapy supplemented with S. boulardii CNCM I-745 (approximately 22.5 x 10^9 CFU) for 14 days.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saccharomyces boulardii (Experimental): Conventional treatment (amoxicillin 1 g three times a day, tinidazole 1g four times a day, and omeprazole 40mg twice a day; n=34) plus S. boulardii CNCM I-745 (approximately 22.5 x109 CFU
  Interventions: Drug: Saccharomyces Boulardii-Containing Product in Oral Dose Form
- No intervention (No Intervention): Conventional treatment (amoxicillin 1 g three times a day, tinidazole 1g four times a day, and omeprazole 40mg twice a day; n=34)

INTERVENTIONS:
Drug: Saccharomyces Boulardii-Containing Product in Oral Dose Form — S. boulardii CNCM I-745 (approximately 22.5 x109 CFU)
  Arms: Saccharomyces boulardii

SUMMARY:
Eradication therapy against Helicobacter pylori (Hp) carries adverse effects, such as altering the intestinal microbiota's structure and function and selecting commensals and pathogens resistant to antibiotics. This last undesirable effect turns the microbiota into a reservoir of resistance genes. Saccharomyces boulardii CNCM I-745 (Sb) can improve dysbiosis and reduce the abundance of multi-resistant bacteria. The objective of the current project is to characterize the resistome of individuals treated with anti-H. pylori therapy in the presence or absence of Sb in fecal samples. Applying metagenomics and using next-generation sequencing tools, the investigators seek to demonstrate the beneficial effect of Sb on the gut microbiota by reducing the abundance of resistance genes and characterizing bacteria modulated by this probiotic-yeast. The investigators expect to find an increase in the diversity and relative abundance of antibiotic resistance genes (ARGs) in the intestine of participants who did not receive Sb during Hp eradication therapy and one month after completing treatment. The increase in ARGs is probably correlated with the presence of Clostridia and Bacteroides.

DETAILED DESCRIPTION:
Antibiotic use is one of the most common therapeutic strategies of modern medicine. Together with the significant beneficial effects of antibiotic use, side effects accompany the use of these drugs, including the increasing appearance of antibiotic-resistant microbes, a global public health problem. Other significant side effects include gastrointestinal-related symptoms such as diarrhea, pain, intestinal discomfort, and flatulence, which can be the consequence of dysbiosis. A common strategy to limit antibiotic-associated side effects is the addition of probiotics, as S. boulardii CNCM I-745 (Sb). The use of bacterial probiotics to reduce antibiotic-associated side effects has several potential limitations, including the destruction of probiotics, development of probiotics strains resistant to antibiotics, and passage of antibiotic-resistant genes to pathogenic bacteria through horizontal gene transfer. Sb is a probiotic yeast whose benefits on intestinal dysbiosis have been associated with establishing a favorable growth environment for the normal intestinal microbiota. Due to the yeast nature of this probiotic, the limitations of bacterial-probiotics cannot be accounted for during Sb use. Consequently, it is crucial to study the molecular mechanism elicited by Sb on intestinal microbiota, including changes in resistome.

In our previous study regarding the supplementation with Sb on the treatment against H. pylori (Hp) infection, patients that received the probiotic had a significantly lower frequency of gastrointestinal symptoms. Additionally, those patients have a higher number of bacterial diversity evenness (P=0.0156), higher abundance of Enterobactereacea, and lower abundance of Bacteroides and Clostridia upon treatment completion and one month later. Bacteroides and Clostridia have been previously implicated as antibiotic multi-resistant pro-inflammatory strains. The objective of the current project is to characterize the resistome of individuals treated with anti-H. pylori therapy in the presence or absence of Sb in fecal samples.

Specific aims To determine the resistome changes before and after Hp eradication treatment in patients that have received or not Sb.

To compare the resistome patterns between patients treated for Hp infection that have received or not SB, at the time of completion of treatment and one month after finishing them.

Based on the shotgun metagenomics, the researchers seek to characterize the microbiome and resistome in fecal samples and understand the microbiome's functional characteristics, including virulence genes, metabolic pathways, and mobile genetic elements.

Methodology DNA obtained from the previous microbiome characterization will be used in this project. In case DNA is not enough, the researchers will extract DNA from the frozen stored samples using the Power Soil kit.

DNA will be shipped to UNC Chapel Hill or the University of Minnesota, where genomic libraries will be constructed. Hi-Seq Illumina runs will be used to produce a sequencing deepness of 10 million per sample.

FASTQC will be used for reads quality control and multiQC as reports generator from the raw reads. Trimmomatic will be used to trim Illumina adapters and to cut reads on the average quality. As human DNA is present on the fecal samples, the investigators have to remove the host DNA using the mapping software BWA and SAMtools. Using the Resfinder database, the investigators must align the filtered reads and generate a count table using ResistomeAnalyzer. Finally, the researchers can create rarefaction curves based on the table made using AMRPlusPlus.

Expected results The researchers expect to find a higher diversity and abundance of antibiotic resistance genes (genome intrinsic and carried by mobile genetic elements) on the group that did not receive Sb at the end of treatment and one month after its completion. This would be correlated with the lower abundance of Clostridia and Bacteroides encountered in the 16S rRNA gene microbiome characterization.

The investigators will also be able to sub-characterize the resistome diversity and abundance of antibiotic resistance genes encountered typically on Enterobacteriaceae. A previous analysis found a higher abundance of Enterobacteriaceae in the group that received Sb (previously reported in a mouse model by Sovran et al. 2018). Additionally, since the researchers will obtain the raw reads on the shotgun sequencing, they could further characterize the bacteria modulated by the use of Sb at strain level (Bacteroides, Clostridia, and Enterobacteriaceae). Together, the researchers expect to obtain valuable data on the use of Sb regarding antibiotic resistance and further microbiome characteristics, including genes of bacterial pathogenicity. These results will contribute to clarify the beneficial effects of Sb addition in patients treated for Hp infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with typical dyspepsia symptoms from whom an upper gastrointestinal endoscopy with biopsies was done for histopathological examination.

Exclusion Criteria:

* Pregnancy or lactation.
* Subjects diagnosed with another gastrointestinal disease such as inflammatory bowel disease and malabsorption syndromes.
* Subjects taking or are planning to take pre- pro- or symbiotic.
* Subjects that have received antibiotics in the last month for any reason.
* Subjects who have received corticosteroids chronically for any reason; have received medication to inhibit nutrient absorption; use of NSAID during the last month that cannot stop the treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2017-06-09 (Actual)

PRIMARY OUTCOMES:
Modifications in the fecal resistome during a probiotic administration | Participating patients were asked to provide three fecal samples during the study, the first before initiation of antibiotics, the second immediately after completion of antibiotics, and the last sample 1 month after finishing the treatment.
  Changes in abundance and diversity of antimicrobial resistance genes in fecal micobiota from individuals treated against a H. pylori infection with Saccharomyces boulardii CNCM I-745 as an additional therapy to conventional treatment regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Paúl A Cárdenas, PhD, Principal Investigator — Universidad San Francisco de Quito

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (DNA sequences).
Time Frame: DNA sequences (raw reads): immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Background] Cardenas PA, Garces D, Prado-Vivar B, Flores N, Fornasini M, Cohen H, Salvador I, Cargua O, Baldeon ME. Effect of Saccharomyces boulardii CNCM I-745 as complementary treatment of Helicobacter pylori infection on gut microbiome. Eur J Clin Microbiol Infect Dis. 2020 Jul;39(7):1365-1372. doi: 10.1007/s10096-020-03854-3. Epub 2020 Mar 3. PMID 32125555
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32125555/